CLINICAL TRIAL: NCT05119946
Title: A Pilot Study of the Effectiveness of a Suicide Prevention Video Tool to Reduce the Incidence of Active Suicide Behavior in Individuals With Psychiatric Illness
Brief Title: A Feasibility Study of a Suicide Prevention Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHREB 2015-141
Record Dates: First submitted 2016-08-23; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Suicidal Ideation; Suicide Attempts; Psychiatric Illness
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suicide prevention video (Experimental): In this group, in addition to receiving the standard of care for their suicidality, the participants will also view a suicide prevention video.
  Interventions: Behavioral: Suicide prevention video; Other: Standard suicide treatment
- Standard suicide treatment (Active Comparator): In this group, participants will only receive the standard of care for their suicidality, which can include medications and/or therapy. The care will be determine by their attending physician.
  Interventions: Other: Standard suicide treatment

INTERVENTIONS:
Behavioral: Suicide prevention video — The video has been developed by the research team as an educational tool to teach patients about suicide, the consequences of such and imparting a message of hope.
  Arms: Suicide prevention video
Other: Standard suicide treatment — The standard suicide treatment will be determine by the attending physician and can include medications and/or psychotherapy

SUMMARY:
This initial study is a pilot feasibility study with a primary objective of assessing the feasibility of a larger study by evaluating the procedures and methodology, as well as collecting pilot data. The eventual research goal is to demonstrate whether a suicide prevention video in addition to standard care for suicidality is an effective strategy to reduce suicidal behaviours in individuals with a history of such. The suicide prevention video is developed as an educational tool to inform participants of the various consequences of suicide as well as giving a message of hope. It is hoped that such an approach will help to reduce future suicidal behaviours in those who have a history of such. If so, then this could be made as a part of the standard of care in treating patients with suicidality.

DETAILED DESCRIPTION:
This pilot study will assess the study procedures and methodology to determine the feasibility of a larger study that will be done to asses for any difference in suicidal behaviours when the suicide prevention video is used in addition to standard of care. As such, the primary objectives will include:

* Testing of recruitment, retention, consent, and assignment procedures
* Validating the inclusion/exclusion criteria
* Determining the acceptability and safety of the proposed intervention
* Evaluating implementation procedures and methodology for the intervention
* Evaluating the appropriateness of timing and frequency of data collection points
* Evaluating the appropriateness and feasibility of the assessment tools
* Obtaining parameters for sample size estimation for the larger study
* Assessing the effectiveness of the video medium, content in the video and length of the video

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Admitted to the Royal Columbian Hospital under psychiatric services
* Individuals will have had suicidal behaviours as part of their presentation leading to hospitalization
* Individuals must be at the level 2 observation privileges or higher
* Individuals must be capable of giving consent to participate in the study
* Individuals must speak and read English fluently Individuals admitted to the hospital as voluntary and involuntary (certified) patients

Exclusion Criteria:

* Individuals with hearing or visual deficits that impairs hearing or viewing the SPV
* Individuals who are under the influence of drugs, such as intoxication or active withdrawal
* Individuals with established diagnoses of cognitive impairment affecting their ability to give consent, understand what is expected of them in the study or follow directions
* Patients that require a substitute decision makers to provide consent
* Individuals whose behaviors an/or cognition are actively affected by ongoing psychosis, including hallucinations, delusions, and disorganized behaviors
* Individuals whose treating team assess them as likely to have a negative response to the SPV, for example paranoia around electronic devices
* Patient's who's attending physiatrist is one of the study team members
* Patients who are currently under the direct care of any of the investigators Patients that had acute suicidality in the last 24 hours

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
An assessment of suicidal behaviours following the use of a video intervention | 12 months
  To assess the change in suicidality of patients admitted for such using the Modified Scale for Suicidal Ideation after being given an educational video explaining common misinformation about suicide.

SECONDARY OUTCOMES:
Mean change from baseline in the expression of suicidal ideation on the Modified Scale for Suicidal Ideation at 48 hours, 3 months and 6 months | 12 months
  To measure the change in suicidal behaviours after viewing the video using the "The Modified Scale for Suicidal Ideation". The scale is used to assess the presence or absence of suicide ideation and the degree of severity of suicidal ideas. The benefit of this scale is that it was developed so that paraprofessionals could administer the scale, yet demonstrated excellent internal consistency and interrater reliability, correlated highly with clinician's ratings of suicidal ideation and risk, and discriminated between suicide attempters and nonattempters prior to hospitalization. The scale would be administered at baseline, after watching the video and at 3 and 6 months after watching the video. Each question is scored for a total score that is interpreted as degree of suicidal ideation. Total score range is 0 to 54. Higher scores indicate more severe suicidal ideations. Changes in the total scores will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Hem Phaterpekar, MD, Principal Investigator — Fraser Health
Locations (1):
- Royal Columbian and Eagle Ridge Hospitals, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No